CLINICAL TRIAL: NCT06443632
Title: WASPE Sleep Adjustment for Children Aged 0-4 Years Undergoing Radiation Therapy: A Prospective Randomized Controlled Phase II Clinical Trial
Brief Title: WASPE Sleep Adjustment for Children Aged 0-4 Years Undergoing Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Director of Radiation Oncology Department, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SDZLEC2024-077-01
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Cancer
Keywords: Pediatric cancer; Radiotherapy; Sleep adjustment
MeSH Terms: conditions — Neoplasms | interventions — Chloral Hydrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WASPE Sleep Adjustment Protocol (Experimental): Parents are instructed to implement the WASPE protocol (Watching videos, Activities outdoors, Stimulation to stay awake, Playing with toys, and Eating snacks) to keep the child awake from morning until the scheduled RT slot (14:00-16:00), thereby inducing natural deep sleep during RT without pharmacologic sedation. Treatment setup is verified with CBCT and monitored in real time using OSMS with a 5-mm motion threshold.
  Interventions: Behavioral: WASPE Sleep Adjustment Protocol
- Sedation (Active Comparator): Oral or rectal chloral hydrate (typically 30-50 mg/kg, maximum 1 g) administered approximately 30 minutes before each RT fraction per institutional pediatric sedation protocol. Vital signs are monitored continuously. CBCT and OSMS are used as in the experimental arm.
  Interventions: Drug: Chloral Hydrate

INTERVENTIONS:
Behavioral: WASPE Sleep Adjustment Protocol — Parents are instructed to implement the WASPE protocol (Watching videos, Activities outdoors, Stimulation to stay awake, Playing with toys, and Eating snacks) to keep the child awake from morning until the scheduled RT slot (14:00-16:00), thereby inducing natural deep sleep during RT without pharmacologic sedation. Treatment setup is verified with CBCT and monitored in real time using OSMS with a 5-mm motion threshold.
  Arms: WASPE Sleep Adjustment Protocol
Drug: Chloral Hydrate — Oral or rectal chloral hydrate (typically 30-50 mg/kg, maximum 1 g) administered approximately 30 minutes before each RT fraction per institutional pediatric sedation protocol. Vital signs are monitored continuously. CBCT and OSMS are used as in the experimental arm.
  Arms: Sedation

SUMMARY:
This prospective, randomized controlled feasibility trial aims to evaluate the feasibility and effectiveness of a behavioral sleep adjustment protocol (WASPE: Watching videos, Activities outdoors, Stimulation to stay awake, Playing with toys, Eating snacks) in pediatric patients undergoing radiotherapy. A total of 48 children aged 0-4 years with non-head-and-neck tumors were enrolled and allocated to either the WASPE sleep adjustment group or the sedation group. The primary outcome was the rate of radiotherapy completion without sedation in the WASPE group. Secondary outcomes included motion accuracy (CBCT and OSMS) and physiological biomarkers (IgA, IgG, IgM, GH). This study explores a non-pharmacological alternative to sedation in pediatric radiotherapy preparation.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, pragmatic feasibility trial comparing a structured behavioral sleep-adjustment protocol (WASPE) with standard pharmacologic sedation to support radiotherapy (RT) delivery in children 0-4 years. Eligible patients have non-head-and-neck solid tumors indicated for external-beam RT and are randomized 2:1 to WASPE or sedation. To focus on children who typically require assistance to complete daily RT, those able to maintain treatment position without assistance are excluded.

The WASPE workflow is caregiver-guided and begins ≥3 days before RT to build sleep pressure: early wake (≈06:00-07:00), late bedtime (≈22:00-23:00), and RT scheduled 14:00-16:00 to coincide with a natural nap; familiarization with the treatment environment is encouraged. During treatment, motion is monitored with an optical surface monitoring system (OSMS) using a 5-mm threshold; if deviation exceeds the threshold and does not self-correct, irradiation is paused, the child is repositioned, and alignment is re-verified with CBCT. The control arm receives chloral hydrate 30-50 mg/kg (max 1 g) orally or rectally ~30 minutes before treatment per institutional protocol with continuous cardiorespiratory monitoring. Rescue sedation may be used as medically necessary and is recorded; caregiver-requested crossover from the sedation arm to WASPE is permitted.

Pre-treatment CBCT is registered to the planning CT at each fraction to correct set-up error. Real-time surface tracking is performed with OSMS.

The primary outcome is the per-fraction sedation-free completion rate in the WASPE arm, evaluated for non-inferiority to a prespecified performance target (95% with a 2% margin; lower 95% CI > 93%). Secondary outcomes include inter- and intrafraction displacement (CBCT/OSMS), serum IgA/IgG/IgM and growth hormone measured ≤3 days before RT and ≈7 days after completion, and safety per CTCAE v5.0 (including treatment interruptions and rescue sedation).

ELIGIBILITY:
Inclusion Criteria:

* Age 0-4 years, any sex.
* Histologically confirmed malignant solid tumor indicated for external-beam radiotherapy.
* Lansky performance status ≥ 70.
* Expected survival ≥ 3 months.
* Adequate organ function within 14 days prior to enrollment, as determined by the investigator.
* Parent(s)/legal guardian(s) able and willing to follow the WASPE instructions and provide written informed consent.
* Clinical expectation that pharmacologic sedation or a structured behavioral intervention (e.g., WASPE) would otherwise be needed to complete radiotherapy.

Exclusion Criteria:

* Ability to maintain treatment position without assistance (i.e., child already tolerates RT without sedation/behavioral intervention).
* Head and neck tumors requiring thermoplastic mask immobilization incompatible with OSMS in our workflow.
* Sleep disorders or central nervous system dysfunction affecting sleep-wake regulation or protocol compliance.
* Clinically significant growth retardation or immunologic impairment judged by the investigator.
* Severe or uncontrolled systemic disease or infection that could interfere with participation.
* Contraindication or known allergy to chloral hydrate.
* Any other condition that, in the investigator's judgment, would preclude safe participation or reliable assessment of outcomes.

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Per-fraction radiotherapy completion without pharmacologic sedation (WASPE arm) | From the first radiotherapy fraction through completion of the radiotherapy course (all scheduled fractions), with final assessment at the end of radiotherapy (typically within 2-8 weeks from treatment initiation).
  A fraction is counted successful if completed as planned without rescue sedation. The primary analysis evaluates non-inferiority to a prespecified performance target of 95% with a 2% margin; non-inferiority is concluded if the lower bound of the 95% CI exceeds 93.0% (one-sided α = 0.025). Fractions are analyzed under an intention-to-treat framework at the fraction level.

SECONDARY OUTCOMES:
Radiotherapy positioning accuracy (CBCT/OSMS) | From the first radiotherapy fraction through completion of the radiotherapy course, with final assessment at the end of radiotherapy (typically within 2-8 weeks from treatment initiation).
  Interfraction setup error is quantified using pre-treatment CBCT registration to the planning CT along lateral, longitudinal, and vertical axes. Intrafraction motion is assessed using real-time optical surface monitoring system (OSMS) tracking, including total deviation and beam-on deviation metrics. A 5-mm motion threshold is applied; persistent deviations trigger treatment pause, patient repositioning, and CBCT re-verification as clinically indicated.
Serum immunoglobulins (IgA, IgG, IgM) | ≤ 3 days before radiotherapy and ≈ 7 days after completion
  Peripheral blood samples analyzed by ELISA to quantify IgA/IgG/IgM; change from pre-RT to post-RT compared between groups.
Serum growth hormone (GH) | ≤ 3 days before radiotherapy and ≈ 7 days after completion
  Serum GH measured by chemiluminescent immunoassay; change from pre-RT to post-RT compared between groups.
Safety (CTCAE v5.0) | During radiotherapy and ≈ 7 days post-RT
  Incidence and severity of AEs/SAEs graded per CTCAE v5.0, plus treatment interruptions and rescue sedation use.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Dorcter, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Department of Radiation Oncology, Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bhakta N, Force LM, Allemani C, Atun R, Bray F, Coleman MP, Steliarova-Foucher E, Frazier AL, Robison LL, Rodriguez-Galindo C, Fitzmaurice C. Childhood cancer burden: a review of global estimates. Lancet Oncol. 2019 Jan;20(1):e42-e53. doi: 10.1016/S1470-2045(18)30761-7. PMID 30614477
- [Result] Ni X, Li Z, Li X, Zhang X, Bai G, Liu Y, Zheng R, Zhang Y, Xu X, Liu Y, Jia C, Wang H, Ma X, Zheng H, Su Y, Ge M, Zeng Q, Wang S, Zhao J, Zeng Y, Feng G, Xi Y, Deng Z, Guo Y, Yang Z, Zhang J. Socioeconomic inequalities in cancer incidence and access to health services among children and adolescents in China: a cross-sectional study. Lancet. 2022 Sep 24;400(10357):1020-1032. doi: 10.1016/S0140-6736(22)01541-0. PMID 36154677
- [Result] Jairam V, Roberts KB, Yu JB. Historical trends in the use of radiation therapy for pediatric cancers: 1973-2008. Int J Radiat Oncol Biol Phys. 2013 Mar 1;85(3):e151-5. doi: 10.1016/j.ijrobp.2012.10.007. Epub 2012 Dec 27. PMID 23273995
- [Result] McMullen KP, Hanson T, Bratton J, Johnstone PA. Parameters of anesthesia/sedation in children receiving radiotherapy. Radiat Oncol. 2015 Mar 11;10:65. doi: 10.1186/s13014-015-0363-2. PMID 25889312
- [Result] Yildirim I, I Celik A, B Bay S, Pasin O, Tutuncu AC. Propofol-based balanced anesthesia is safer in pediatric radiotherapy. J Oncol Pharm Pract. 2019 Dec;25(8):1891-1896. doi: 10.1177/1078155218825296. Epub 2019 Jan 30. PMID 30700212
- [Result] Cote CJ, Wilson S. Guidelines for Monitoring and Management of Pediatric Patients Before, During, and After Sedation for Diagnostic and Therapeutic Procedures. Pediatr Dent. 2019 Jul 15;41(4):259-260. PMID 31439084
- [Result] Stratmann G, Sall JW, May LD, Bell JS, Magnusson KR, Rau V, Visrodia KH, Alvi RS, Ku B, Lee MT, Dai R. Isoflurane differentially affects neurogenesis and long-term neurocognitive function in 60-day-old and 7-day-old rats. Anesthesiology. 2009 Apr;110(4):834-48. doi: 10.1097/ALN.0b013e31819c463d. PMID 19293705
- [Result] Briner A, De Roo M, Dayer A, Muller D, Habre W, Vutskits L. Volatile anesthetics rapidly increase dendritic spine density in the rat medial prefrontal cortex during synaptogenesis. Anesthesiology. 2010 Mar;112(3):546-56. doi: 10.1097/ALN.0b013e3181cd7942. PMID 20124985
- [Result] Haeberli S, Grotzer MA, Niggli FK, Landolt MA, Linsenmeier C, Ammann RA, Bodmer N. A psychoeducational intervention reduces the need for anesthesia during radiotherapy for young childhood cancer patients. Radiat Oncol. 2008 Jun 4;3:17. doi: 10.1186/1748-717X-3-17. PMID 18522761
- [Result] Gutkin PM, Skinner L, Jiang A, Donaldson SS, Loo BW Jr, Oh J, Wang YP, von Eyben R, Snyder J, Bredfeldt JS, Breneman JC, Constine LS, Faught AM, Haas-Kogan D, Holmes JA, Krasin M, Larkin C, Marcus KJ, Maxim PG, McClelland S 3rd, Murphy B, Palmer JD, Perkins SM, Shen CJ, Terezakis S, Bush K, Hiniker SM. Feasibility of the Audio-Visual Assisted Therapeutic Ambience in Radiotherapy (AVATAR) System for Anesthesia Avoidance in Pediatric Patients: A Multicenter Trial. Int J Radiat Oncol Biol Phys. 2023 Sep 1;117(1):96-104. doi: 10.1016/j.ijrobp.2023.03.063. Epub 2023 Mar 30. PMID 37001762
- [Result] Liu P, Huang Q, Zhang T, Zhang X, Shi P, Qi L, Yue J. WASPE Sleep Deprivation, Paired with an Optical Surface Monitoring System, Can Provide Accurate Radiation Therapy to Pediatric Patients Without the Need for Sedation. Pract Radiat Oncol. 2023 May-Jun;13(3):e292-e300. doi: 10.1016/j.prro.2022.11.007. Epub 2022 Dec 6. PMID 36494032
- [Result] Lawler G. A review of surface guidance in extracranial stereotactic body radiotherapy (SBRT/SABR) for set-up and intra-fraction motion management. Tech Innov Patient Support Radiat Oncol. 2022 Jan 19;21:23-26. doi: 10.1016/j.tipsro.2022.01.001. eCollection 2022 Mar. PMID 35079644
- [Result] Varni JW, Burwinkle TM, Katz ER, Meeske K, Dickinson P. The PedsQL in pediatric cancer: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales, Multidimensional Fatigue Scale, and Cancer Module. Cancer. 2002 Apr 1;94(7):2090-106. doi: 10.1002/cncr.10428. PMID 11932914
- [Result] Dunstan DA, Scott N. Norms for Zung's Self-rating Anxiety Scale. BMC Psychiatry. 2020 Feb 28;20(1):90. doi: 10.1186/s12888-019-2427-6. PMID 32111187